CLINICAL TRIAL: NCT04672837
Title: Efficacy of Pediatric Integrative Manual Therapy in Babies With Deformational Plagiocephaly and Congenital Muscular Torticollis
Brief Title: Pediatric Integrative Manual Therapy in Babies With Deformational Plagiocephaly and Congenital Muscular Torticollis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Iñaki Pastor Pons, Principal Investigator at Manual Therapy Research Unit, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PMT2
Record Dates: First submitted 2020-12-02; First posted 2020-12-17 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Plagiocephaly, Nonsynostotic; Plagiocephaly, Positional; Congenital Muscular Torticollis
Keywords: Manual Therapy; Physical Therapy; Cranial Asymmetry; Preferential position of the head
MeSH Terms: conditions — Plagiocephaly, Nonsynostotic; Congenital torticollis

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double (Investigator, Outcomes Assessor) The assessors who receive participants and do the measurement are masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Therapy Group (Experimental): 10 sessions of Pediatric Manual Therapy, once a week. Soft cervical mobilisation, myofascial induction and cranial techniques will be administered. Educational physiotherapy consists in "tummy time" stimulation, visual and kinaesthetic stimulation on the non preferential head position and counter position will be also administered.
  Interventions: Procedure: Pediatric Integrative Manual Therapy and educational therapy
- Stretching Group (Active Comparator): A protocol of Stretching at home. 3-5 sessions twice a day. Each stretch will be maintain10 to 30 seconds. Each session 15 will take no less than 15 minutes. 7 days a week.
  Educational Physical Therapy consists in "tummy time" stimulation, visual and kinaesthetic stimulation on the non preferential head position and counter position will be administered.
  Interventions: Procedure: Stretching and educational therapy

INTERVENTIONS:
Procedure: Pediatric Integrative Manual Therapy and educational therapy — Pediatric Integrative Manual Therapy is a soft Orthopedic Manual Therapy approach por infants and children. It integrates joints soft mobilisation, myofascial release and neurodynamic mobilisation. Also the educational therapy.
  Arms: Manual Therapy Group
Procedure: Stretching and educational therapy — It is a protocol of stretching based on literature research. Also the educational therapy with counter positioning, stimulation in prone position, positional care, etc.
  Arms: Stretching Group

SUMMARY:
This study evaluates the efficacy of Pediatric Integrative Manual Therapy in the treatment of positional plagiocephaly in infants. 25 participants will receive a protocol of Pediatric Integrative Manual Therapy and educational physiotherapy in combination, while the other 25 will receive a stretching protocol and educational physiotherapy

DETAILED DESCRIPTION:
The Manual Therapy has shown efficacy in different pathologies in the adult but it is not know its utility in infants and children population, nor in specific pathologies as non synostotic plagiocephaly.

In the conservative treatment of plagiocephaly the educational physiotherapy and the helmet therapy have the better level of evidence among other treatments. When babies present preferential position of the head or Congenital Muscular Torticollis, stretching has shown efficacy.

A protocol of ten sessions of Pediatric Manual Therapy will be applied to infants with positional plagiocephaly in combination with educational physiotherapy. The protocol consists in soft cervical mobilisation, myofascial induction and the application of some pressures to the cranial bones to improve the asymmetry of the head. Educational therapy which consists in more "tummy time" stimulation, stimulation to the non preference position of the head and counter positioning. The control group will receive a protocol of stretching at home done by their parents and Educational therapy.

ELIGIBILITY:
Inclusion Criteria:

* Sign of positional plagiocephaly
* Infants below 12 moths age

Exclusion Criteria:

* No neurological disorders
* No infectious diseases
* No respiratory diseases
* No other treatments

Ages: 0 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Right Oblique Cranial Vault Diameter | 4 weeks
  Measured with caliper, is the distance from left external part of the orbit to the right lambdoid suture at the horizontal plane
Right Oblique Cranial Vault Diameter | 10 weeks
  Measured with caliper, is the distance from left external part of the orbit to the right lambdoid suture at the horizontal plane
Left Oblique Cranial Vault Diameter | 4 weeks
  Measured with caliper, is the distance from right external part of the orbit to the left lambdoid suture at the horizontal plane
Left Oblique Cranial Vault Diameter | 10 weeks
  Measured with caliper, is the distance from right external part of the orbit to the left lambdoid suture at the horizontal plane
Active Cervical Rotation Range of movement | 4 weeks
  Measured with photographs and digital angular analysis
Active Cervical Rotation Range of movement | 10 weeks
  Measured with digital angular analysis
Passive Cervical Rotation Range of movement | 4 weeks
  Measured lying down with joint goniometer
Passive Cervical Rotation Range of movement | 10 weeks
  Measured lying down with joint goniometer
Passive Cervical Lateral Flexion Range of movement | 4 weeks
  Measured lying down with joint goniometer
Passive Cervical Lateral Flexion Range of movement | 10 weeks
  Measured lying down with joint goniometer
Muscle Function Test | 4 weeks
  Measured in lateral suspension giving a value of 0 to 5 according to the alignment of the head with the trunk
Muscle Function Test | 10 weeks
  Measured in lateral suspension giving a value of 0 to 5 according to the alignment of the head with the trunk

SECONDARY OUTCOMES:
Cranial length | 4 weeks and 10 weeks
  Measured with calliper, is the distance from most anterior point in the frontal bone in the middle line to the most posterior point in the cranial vault on the horizontal plane in the middle line
Cranial length | 10 weeks
  Measured with calliper, is the distance from most anterior point in the frontal bone in the middle line to the most posterior point in the cranial vault on the horizontal plane in the middle line
Cranial wide | 4 weeks
  Measured with calliper, is the distance between the two more lateral points in the vault, usually in the temporal or parietal bone.
Cranial wide | 10 weeks
  Measured with calliper, is the distance between the two more lateral points in the vault, usually in the temporal or parietal bone.
Cranial maximal circumference | 4 weeks
  Measured in cm with a measuring tape.
Cranial maximal circumference | 10 weeks
  Measured in cm with a measuring tape.
Alberta Infant Motor Scale | 10 weeks
  Neuromotor scale for infants from 0 to 14 months. Maximum value 90th; minimum value 0th. Higher scores indicate a better motor and postural development. Values below 15th indicate risk of development delay.
Visual Analogical Scale about improvement in cervical movement after intervention | 10 weeks
  Parents perception of changes in their baby. Minimum value -10; maximum value +10. Higher scores indicate a better perception of change in the cervical movement.
Visual Analogical Scale about improvement in cranial asymmetry after intervention | 10 weeks
  Parents perception of changes in their baby. Minimum value -10; maximum value +10. Higher scores indicate a better perception of change in the head shape

CONTACTS AND LOCATIONS:
Overall Officials: Orosia Lucha, Study Chair — Universidad de Zaragoza
Locations (1):
- Instituto deTerapias Integrativas, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Billi M, Greco A, Colonneli P, Volpi G, Valente D, Galeoto G. The functional manual therapy intervention in infants with non-synostotic plagiocephaly: a pilot study. Minerva Pediatr (Torino). 2022 Jun;74(3):294-300. doi: 10.23736/S2724-5276.17.04838-1. Epub 2017 Oct 25. PMID 29072040
- [Background] Cabrera-Martos I, Valenza MC, Valenza-Demet G, Benitez-Feliponi A, Robles-Vizcaino C, Ruiz-Extremera A. Effects of manual therapy on treatment duration and motor development in infants with severe nonsynostotic plagiocephaly: a randomised controlled pilot study. Childs Nerv Syst. 2016 Nov;32(11):2211-2217. doi: 10.1007/s00381-016-3200-5. Epub 2016 Jul 27. PMID 27465676
- [Background] Bagagiolo D, Didio A, Sbarbaro M, Priolo CG, Borro T, Farina D. Osteopathic Manipulative Treatment in Pediatric and Neonatal Patients and Disorders: Clinical Considerations and Updated Review of the Existing Literature. Am J Perinatol. 2016 Sep;33(11):1050-4. doi: 10.1055/s-0036-1586113. Epub 2016 Sep 7. PMID 27603533
- [Background] Ballardini E, Sisti M, Basaglia N, Benedetto M, Baldan A, Borgna-Pignatti C, Garani G. Prevalence and characteristics of positional plagiocephaly in healthy full-term infants at 8-12 weeks of life. Eur J Pediatr. 2018 Oct;177(10):1547-1554. doi: 10.1007/s00431-018-3212-0. Epub 2018 Jul 20. PMID 30030600
- [Background] Williams E. Preventing "Flat-headed" Babies: A Commentary on "Impact of Parent Practices of Infant Positioning on Head Orientation Profile and Development of Positional Plagiocephaly in Healthy Term Infants". Phys Occup Ther Pediatr. 2018 Feb;38(1):15-17. doi: 10.1080/01942638.2018.1405661. No abstract available. PMID 29372872
- [Background] Nahles S, Klein M, Yacoub A, Neyer J. Evaluation of positional plagiocephaly: Conventional anthropometric measurement versus laser scanning method. J Craniomaxillofac Surg. 2018 Jan;46(1):11-21. doi: 10.1016/j.jcms.2017.10.010. Epub 2017 Oct 16. PMID 29137851
- [Background] van Vlimmeren LA, Engelbert RH, Pelsma M, Groenewoud HM, Boere-Boonekamp MM, der Sanden MW. The course of skull deformation from birth to 5 years of age: a prospective cohort study. Eur J Pediatr. 2017 Jan;176(1):11-21. doi: 10.1007/s00431-016-2800-0. Epub 2016 Nov 4. PMID 27815732
- [Background] Aarnivala H, Vuollo V, Harila V, Heikkinen T, Pirttiniemi P, Valkama AM. Preventing deformational plagiocephaly through parent guidance: a randomized, controlled trial. Eur J Pediatr. 2015 Sep;174(9):1197-208. doi: 10.1007/s00431-015-2520-x. Epub 2015 Apr 1. PMID 25823758
- [Background] De Bock F, Braun V, Renz-Polster H. Deformational plagiocephaly in normal infants: a systematic review of causes and hypotheses. Arch Dis Child. 2017 Jun;102(6):535-542. doi: 10.1136/archdischild-2016-312018. Epub 2017 Jan 19. PMID 28104626
- [Background] Ohman A, Mardbrink EL, Stensby J, Beckung E. Evaluation of treatment strategies for muscle function in infants with congenital muscular torticollis. Physiother Theory Pract. 2011 Oct;27(7):463-70. doi: 10.3109/09593985.2010.536305. Epub 2011 May 15. PMID 21568831
- [Background] Ohman A, Nilsson S, Beckung E. Stretching treatment for infants with congenital muscular torticollis: physiotherapist or parents? A randomized pilot study. PM R. 2010 Dec;2(12):1073-9. doi: 10.1016/j.pmrj.2010.08.008. PMID 21145518
- [Background] Ohman AM, Nilsson S, Beckung ER. Validity and reliability of the muscle function scale, aimed to assess the lateral flexors of the neck in infants. Physiother Theory Pract. 2009 Feb;25(2):129-37. doi: 10.1080/09593980802686904. PMID 19212900
- [Background] Di Chiara A, La Rosa E, Ramieri V, Vellone V, Cascone P. Treatment of Deformational Plagiocephaly With Physiotherapy. J Craniofac Surg. 2019 Oct;30(7):2008-2013. doi: 10.1097/SCS.0000000000005665. PMID 31232996
- [Background] Systematic Review and Evidence-Based Guidelines for the Management of Patients with Positional Plagiocephaly. Pediatrics. 2016 Nov;138(5):e20162802. doi: 10.1542/peds.2016-2802. No abstract available. PMID 27940801